CLINICAL TRIAL: NCT05169866
Title: A Randomized Active-Controlled Study Comparing Efficacy and Safety of Nifekalant to Amiodarone in New-Onset Atrial Fibrillation After Cardiac Surgery
Brief Title: Nifekalant Versus Amiodarone in New-Onset Atrial Fibrillation After Cardiac Surgery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Xiaotong Hou, Professor, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-15
Record Dates: First submitted 2021-11-29; First posted 2021-12-27 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: New Onset Atrial Fibrillation; Complications; Cardiac, Postoperative
Keywords: Nifekalant; Amiodarone; Cardiac Surgery; Postoperative Atrial Fibrillation
MeSH Terms: interventions — nifekalant; Amiodarone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous Nifekalant (Experimental): Patients randomized to Nifekalant arm will receive a bolus of 0.3mg/kg IV in the first 5 minutes and a maintenance dose of 0.2-0.4mg/kg/h for 24 hours. If the patient has a recurrence of atrial fibrillation, the maintenance dose can be increased (up to 0.8 mg/kg/h) according to the patient's condition, or receive a bolus of 3mg/kg again at 2 hours intervals. Nifekalant is administered for 24 hours unless meeting the criteria for discontinuation.
  Interventions: Drug: Nifekalant
- Intravenous Amiodarone (Active Comparator): Patients randomized to an amiodarone arm will receive a bolus of 150mg IV in the first 10 minutes and a maintenance dose of 0.5-1mg/min for 24 hours. If the patient has a recurrence of atrial fibrillation, the dosage can be adjusted according to the patient's condition, but the total dosage administered within 24 hours should not exceed 2g. Amiodarone is administered for 24 hours unless meeting the criteria for discontinuation.
  Interventions: Drug: Amiodarone

INTERVENTIONS:
Drug: Nifekalant — Patients identified with new-onset atrial fibrillation with a sustained duration of greater than 1 minutes and less than 48 hours will be considered for the study. Patients randomized to nifekalant arm will receive a bolus of 0.3mg/kg IV in the first 5 minutes and a maintenance dose of 0.2-0.4mg/kg/h for 24 hours.
  Other Names: Nifekalant Hydrochloride
  Arms: Intravenous Nifekalant
Drug: Amiodarone — Patients identified with new-onset atrial fibrillation with a sustained duration of greater than 1 minutes and less than 48 hours will be considered for the study. Patients randomized to amiodarone arm will receive a bolus of 150mg IV in the first 10 minutes and a maintenance dose of 0.5-1mg/min for 24 hours.
  Other Names: Amiodarone Hydrochloride
  Arms: Intravenous Amiodarone

SUMMARY:
Postoperative atrial fibrillation is a major complication of cardiac surgery, which could lead to high morbidity and mortality, increase duration of hospital stay and increase the cost of treatment. New-onset atrial fibrillation after cardiac surgery is considered as a multifactorial phenomenon. Amiodarone, the most commonly used drug for cardioversion, is limited in atrial fibrillation after cardiac surgery due to side effects such as hypotension, bradycardia, and extracardiac side effects. Nifekalant is a novel class III antiarrhythmic agent with short onset time. It is a pure potassium channel blocker, which generally does not cause hypotension and bradycardia. There have been several trials that proven efficacy of nifekalant in converting persistent atrial fibrillation. For atrial fibrillation after cardiac surgery, the effectiveness and safety of nifekalant compared to amiodarone have not yet been reported. The investigators plan to perform a clinical trial comparing nifekalant to amiodarone in new-onset atrial fibrillation after cardiac surgery patients with a primary outcome of cardioversion at 4 hours. Secondary outcomes will follow cardioversion at 90 minutes and 24 hours, maintenance time of sinus rhythm within 24 hours, average time to conversion to sinus rhythm, rate of hypotension, length of ICU stay, length of hospital stay and hospital mortality.

DETAILED DESCRIPTION:
1. Background: Atrial fibrillation (AF) is the most common cardiac arrhythmia post cardiac surgery. Estimates suggest that rates of patients experiencing AF after cardiac surgery exceeds 30%. AF has multiple effects on the cardiopulmonary hemodynamics. New-onset atrial fibrillation after cardiac surgery is considered as a multifactorial phenomenon. Its pathogenesis is characterized by inflammation, oxidative stress and autonomic dysfunction. AF after cardiac surgery could lead to high morbidity and mortality, increase duration of hospital stay and increase the cost of treatment. Treatment of AF include rhythm control and rate control. Typical rate control agents are contraindicated due to need of vasoactive requirements. The 2017 EACTS Guidelines on perioperative medication in adult cardiac surgery recommends that in patients with hemodynamically stable postoperative AF, rhythm control is recommended (I, B). Currently, amiodarone is most commonly used drug for rhythm control. It has long onset and cardioversion time. It can also cause side effects such as hypotension, typically requiring escalating doses of vasoactive medications. Other side effects include bradycardia, and extracardiac side effects in lung, liver and thyroid, which limit the clinical application of amiodarone in AF after cardiac surgery. Nifekalant is a novel class III antiarrhythmic agent with short onset time. It is a pure potassium channel blocker, which generally does not cause hypotension and bradycardia. Nifekalant prolongs the action potential duration and effective refractory period of atrial and ventricular myocytes, and prolong the QT interval. There have been several trials that proven efficacy of nifekalant in converting persistent atrial fibrillation. For new-onset AF post cardiac surgery, the effectiveness and safety of nifekalant compared to standard of care amiodarone have not yet been reported.
2. Research hypothesis: For patients with new-onset atrial fibrillation after cardiac surgery, administration of nifekalant is not inferior to amiodarone in terms of rate of cardioversion to sinus rhythm at 4 hours.
3. Methods: Patients after cardiac surgery will be recruited from the ICU based on inclusion and exclusion criteria. Patients identified with new-onset atrial fibrillation with a sustained duration of greater than 1 minutes and less than 48 hours will be considered for the study. Patients will be randomized to amiodarone versus nifekalant using a computerized process. The primary outcome is rate of cardioversion at 4 hours. Secondary outcomes include rates of cardioversion at 90 minutes and 24 hours, maintenance time of sinus rhythm within 24 hours, average time to cardioversion to sinus rhythm, rate of hypotension, length of ICU stay, length of hospital stay and hospital mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, <85 years old, no gender limit;
2. Postoperative atrial fibrillation in the ICU after cardiac surgery;
3. The duration of atrial fibrillation> 1 minute, and ≤ 48 hours;
4. Hemodynamically stable (no need to increase vasoactive drugs and SBP>90/MAP>60mmHg);
5. After pre-treatment (including: correcting electrolyte disturbances, optimizing volume status, improving oxygenation, controlling body temperature, analgesia and minimizing the use of inotropes and vasopressors), the clinician believes that antiarrhythmic drugs are needed.
6. Obtained the informed consent from the patients or their family members.

Exclusion Criteria:

1. Heart transplantation, left heart assist device (LVAD) or extracorporeal membrane oxygenation (ECMO) treatment;
2. History of atrial fibrillation/atrial flutter and a history of paroxysmal supraventricular tachycardia;
3. Radiofrequency ablation;
4. Rheumatic heart disease;
5. Complex congenital heart disease (with more than two coexisting congenital heart defects);
6. Cardiac tumors;
7. Transcatheter aortic valve implantation (TAVI), transcatheter mitral valve intervention (TMVI), and transcatheter tricuspid valve intervention (TTVI);
8. Contraindications to amiodarone/nifekalant (PR interval>240ms; 2nd or 3rd degree atrioventricular block (AVB); QT>440ms; familial long QT syndrome; Untreated thyroid disease; AST or ALT>2 times the upper limit; liver cirrhosis; interstitial lung disease);
9. Heart rate (HR) <50 beats/min and/or QRS>140ms without a pacemaker;
10. Received amiodarone or nifekalant within 6 weeks before the operation;
11. Pregnant and lactating female patients;
12. Uncorrected hypokalemia (serum potassium <3.5mmol/L) or hypomagnesemia (whole blood/serum magnesium below the lower limit);
13. Chronic renal failure and/or continuous renal replacement therapy (CRRT);
14. Return to OR during ICU stay or readmission to ICU from Cardiac Surgery ward.
15. Other factors not suitable for participating in this study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2022-05-29 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Rate of cardioversion at 4 hours | 4 hours
  Rate of cardioversion of new-onset atrial fibrillation at 4 hours. The rate of cardioversion = the number of patients who meet the cardioversion criteria in the group / the total number of patients in the group × 100%.
  Cardioversion criteria is: atrial fibrillation stops at least once during the 24 hours observation period and lasts for more than 1 minute.

SECONDARY OUTCOMES:
Rate of cardioversion at 90 minutes | 90 minutes
  Rate of cardioversion of new-onset atrial fibrillation at 90minutes. The rate of cardioversion = the number of cases who meet the cardioversion criteria in the group / the total number of cases in the group × 100%.
Rate of cardioversion at 24 hours | 24 hours
  Rate of cardioversion of new-onset atrial fibrillation at 24 hours. The rate of cardioversion = the number of patients who meet the cardioversion criteria in the group / the total number of patients in the group × 100%.
Maintenance time of sinus rhythm within 24 hours | 24 hours
  The total duration of sinus rhythm within 24 hours.
Average time to AF conversion to sinus rhythm | 24 hours
  Average time from administration of drugs to cardioversion to sinus rhythm.
The incidence of hypotension | 24 hours
  "Hypotension" is defined as: SBP <85mmHg for more than 5 minutes or increase of vasoactive drugs. Incidence = number of cases of hypotension / total number of cases in this group × 100%.
Vasoactive Inotropic Score (VIS) at 90 minutes, 4 hours, and 24 hours | 24 hours
  VIS= Dopamine (ug/kg/min) + dobutamine (ug/kg/min) + 100×adrenaline (ug/kg/min) + 50×levosimendan (ug/kg/min) + 10× milrinone (ug/kg/min) + 10000× vasopressin (unit/kg/min) + 100×norepinephrine (ug/kg/min).
Incidence of severe bradycardia, 3rd degree AVB, severe ventricular arrhythmia | 24 hours
  Severe ventricular arrhythmia: polymorphic/persistent ventricular tachycardia, torsade de pointes (Tdp), ventricular fibrillation. Incidence = number of cases of severe bradycardia, 3rd degree AVB, severe ventricular arrhythmia / total number of cases in this group × 100%.
Liver and kidney function within 24 hours | 24 hours
  Indicators of liver function include ALT and AST. Indicator of kidney function is serum creatinine (Scr).
Cardiac function | 24 hours
  Indicator of cardiac function is left ventricular ejection fraction (LVEF) assessed with echocardiography.
Adverse events | 24 hours
  Adverse medical events that occur after a patient receives a drug, but it does not necessarily have a causal relationship with the treatment.
Co-administration of drugs | 24 hours
  Including patients' basic medications and medications co-administrated during research.
Length of ICU stay | up to 6 months
  Days of patients' stay in ICU
Days of hospital stay | up to 6 months
  Days of patients' stay in hospital
Hospital mortality | up to 6 months
  Mortality of patients during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Xiaotong Hou, MD, PhD, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No